CLINICAL TRIAL: NCT02678065
Title: In.Pact Flexion, a Physician Initiated Trial Investigating the Performance of the In.Pact Admiral Drug-eluting Balloon for the Treatment of Popliteal Lesions
Brief Title: In.Pact Flexion, Investigating the Performance of the In.Pact Admiral DEB for Popliteal Lesions
Acronym: INPCTFLEXION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-120524
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- InPact Admiral (Experimental): Patients treated with the InPact Admiral balloon for popliteal lesions
  Interventions: Device: InPact Admiral DEB

INTERVENTIONS:
Device: InPact Admiral DEB

SUMMARY:
The objective of this study is to evaluate the performance of the In.Pact Admiral DEB for the treatment of popliteal lesions in comparison with literature results of stent treatment in popliteal lesions

ELIGIBILITY:
Inclusion Criteria:

* - De novo, restenotic or reoccluded lesion located in the popliteal artery, with or without superficial femoral artery involvement
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Prior to enrollment, the guidewire has crossed target lesion
* Patient is eligible for treatment with the In.Pact Admiral drug-eluting balloon
* The target lesion, visually estimated, has a maximal length of 14 cm and can be categorized as either a type A or B lesion according the TASC II guidelines
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* Target vessel diameter visually estimated is >3.5mm and <7.5 mm
* There is angiographic evidence of at least one vessel-runoff to the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention.

Exclusion Criteria:

* - Presence of another stent in the target vessel that was placed during a previous procedure
* Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
* Previous by-pass surgery in the same limb
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with known hypersensitivity to nickel-titanium
* Patients with uncorrected bleeding disorders
* Aneurysm located at the level of the SFA and/or popliteal artery
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Ipsilateral iliac treatment before the target lesion procedure with a residual stenosis > 30% or ipsilateral iliac treatment conducted after the target lesion procedure
* Use of thrombectomy, atherectomy or laser devices during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Primary Patency at 12 months | 12 months
  defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) at the target lesion and without TLR within 12 months.

SECONDARY OUTCOMES:
Technical success | 1 day post-op
  defined as the ability to cross and dilate the lesion and achieve residual angiographic stenosis no greater than 30%.
Primary Patency at 1 and 6-months | 1 and 6 months
  defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.4) at the target lesion and without TLR within the time of procedure and the given follow-up
Clinical success at 1, 6 and 12-months | 1, 6 and 12 months
  defined as an improvement of Rutherford classification at 1-, 6- and 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification
Serious Adverse Events | up to 12 months
  defined as a clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization
Survival rate | up to 12 months
  all-cause death ratio
Target Lesion Revascularization | up to 12 months
  defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge
Limb Salvage Rate | up to 12 months
  defined as absence of major amputation. Major amputation is defined as amputation at or above the ankle, as opposed to minor amputation, being an amputation at or below metatarsal level, preserving functionality of the foot)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — Flanders Medical Research Program
Locations (4):
- Belgium (4):
  - Imelda Hospital, Bonheiden, Antwerp
  - A.Z. Sint-Blasius, Dendermonde, East-Flanders
  - OLV Aalst, Aalst, Oost-Vlaanderen
  - RZ Heilig Hart Hospital, Tienen

IPD SHARING:
Plan to Share IPD: Undecided